CLINICAL TRIAL: NCT01892553
Title: Effect of Transcranial Direct Current Stimulation (tDCS) on Acutely Induced Dyspnea in Healthy Volunteers : a Pilot Study
Brief Title: Effect of Non Invasive Brain Stimulation on Experimentally Induced Dyspnea (Breathlessness)
Acronym: tDCS-Dyspnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: Adep Assistance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: acutely2012-A00418-35
Record Dates: First submitted 2013-07-01; First posted 2013-07-04 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Dyspnea
Keywords: Dyspnea; Transcranial direct current stimulation (tDCS); Perception
MeSH Terms: conditions — Dyspnea | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- motor/premotor cortex stimulation (Experimental): Active and sham tDCS applied over the motor/premotor cortex
  Interventions: Device: tDCS
- insular cortex stimulation (Experimental): Active and sham tDCS applied over the insular cortex
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Procedure : 3 different sessions of tDCS (listed below) presented in random order, each applied at a different study visit
  * Anodal tDCS: Intensity of 1.25 milliAmperes (mA) during 15 min
  * Cathodal tDCS: Intensity of 1.25 mA during 15 min
  * Sham tDCS (placebo) (1.25 mA maintained only during the first 30 sec of the 15 minutes application)
  Other Names: Eldith DC stimulator (Magstim Company Ltd. UK)

SUMMARY:
Dyspnea is a frequent, mostly unpleasant and long-lasting, but also often undertreated symptom. Transcranial direct current stimulation (tDCS), a new non invasive method to modify brain activation has shown good efficacy in the treatment of pain especially in the clinical context. Given the fact that dyspnea has many common characteristics with pain, especially concerning the brain areas involved in its central processing, we hypothesize that tDCS may also modify the perception of dyspnea. In order to test this, we first shall determine whether tDCS has a significant effect on acutely induced dyspnea in healthy volunteers. In case of promising results of this pilot study, the next step will be the evaluation of the benefit of tDCS in patients with severe dyspnea.

DETAILED DESCRIPTION:
Dyspnea will be induced by breathing through a combination of an external resistive load and a long tube (inducing CO2 rebreathing) (resulting in a sensation of both increased respiratory effort and air hunger). tDCS will be applied during 15 minutes either over the motor/premotor or over the insular cortex (i.e. 2 brain regions that have previously been shown to be involved in dyspnea perception and/or modulation) in 2 parallel groups of healthy subjects. For each study group, the effect of tDCS on dyspnea perception and on respiratory parameters will be compared between 2 active (anodal and cathodal) and a sham tDCS stimulation (placebo).

ELIGIBILITY:
Inclusion Criteria:

* Registered at the National List of persons taking part in clinical research
* Signed consent form
* Subjects of both genders aged of at least 18 years
* Perfect understanding of the instructions and of sensory scaling
* Prior medical examination

Exclusion Criteria:

* Any current or past disease, in particular respiratory, neurological and psychiatric disorders
* Regular use of drugs, especially those having an impact on respiratory, neurological systems (most specifically those with an effect on the central nervous system)
* Unwilling to participate
* Vulnerable people as defined in the provisions relating to biomedical researches and described in the Code of Public Health.
* Unable to cooperate
* Pregnancy or lactation
* No affiliation to a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Effect of active versus sham tDCS on perceived intensity (sensory component) of induced dyspnea | About 90 min (duration of the study visit)
  Change from baseline (before tDCS application) in intensity of experimentally induced dyspnea (in Borg scale scores) at 4 different time points, 1 during and 3 after each of the 3 tDCS applications (anodal, cathodal and sham)

SECONDARY OUTCOMES:
Effect of active versus sham tDCS on perceived unpleasantness (affective component) of induced dyspnea | About 90 min (duration of the study visit)
  Change from baseline (before tDCS application) in unpleasantness of experimentally induced dyspnea (in Borg scale scores) at 4 different time points, 1 during and 3 after each of the 3 tDCS applications (anodal, cathodal and sham)
Effect of active versus sham tDCS on respiratory variables during induced dyspnea | About 90 min (duration of the study visit)
  Change from baseline (before tDCS application) in mouth pressure swings (cm H2O), tidal volume (L), respiratory frequency (cycles/min), minute ventilation (L/min) and end tidal carbon dioxide (PetCO2)(mm Hg) at 4 different time points, 1 during and 3 after each of the 3 tDCS applications (anodal, cathodal and sham)

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDINE PEIFFER, MD PHD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare, Garches, Garches, France